CLINICAL TRIAL: NCT01343667
Title: The Gore FREEDOM Study: GORE Flow Reversal System and GORE Embolic Filter Extension Study for the Ongoing Collection of Patient Outcomes
Brief Title: GORE Flow Reversal System and GORE Embolic Filter Extension Study
Acronym: FREEDOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRS 09-05
Record Dates: First submitted 2011-04-25; First posted 2011-04-28 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Carotid Stenosis; Constriction, Pathologic; Carotid Artery Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases; Pathological Conditions, Anatomical
Keywords: GORE Neuro Protection System; GORE Flow Reversal System; carotid artery stenosis; embolic protection device; reverse flow; proximal occlusion device; GNPS; Parodi; EMPiRE; distal embolization; minimizing risks of CAS; PAES; embolic filter
MeSH Terms: conditions — Carotid Stenosis; Constriction, Pathologic; Carotid Artery Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases; Pathological Conditions, Anatomical | interventions — Embolic Protection Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GFRS EPD (Other): Carotid artery stenting with Gore Flow Reversal System embolic protection device
  Interventions: Device: Gore Flow Reversal System
- GEF EPD (Other): Carotid artery stenting with Gore Embolic Filter embolic protection device
  Interventions: Device: Gore Embolic Filter

INTERVENTIONS:
Device: Gore Flow Reversal System — Embolic protection by the GORE Flow Reversal System during carotid artery angioplasty and stenting
  Other Names: Neuro Protection System; GORE Neuro Protection System; Parodi; NPS; FRS; PAES; proximal protection
  Arms: GFRS EPD
Device: Gore Embolic Filter — Embolic protection by the GORE Embolic Filter during carotid artery angioplasty and stenting
  Other Names: embolic filter; distal protection
  Arms: GEF EPD

SUMMARY:
The objective of this study is to provide an ongoing evaluation of clinical outcomes associated with the GORE Flow Reversal System and the GORE Embolic Filter when used for embolic protection during carotid artery stenting.

DETAILED DESCRIPTION:
Physicians will have the opportunity to select which embolic protection device, the GORE Flow Reversal System or the GORE Embolic Filter, to use during the carotid artery stenting procedure.

This study is not designed to compare study endpoints between the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Patient, or patient's legal representative, is able and willing to provide informed consent.
* Patient must be at least 18 years of age or older.
* Patient will be selected and treated according to the GORE Flow Reversal System Instructions for Use (IFU) or the GORE Embolic Filter IFU.

Exclusion Criteria:

* Patient is contraindicated for the embolic protection device arm they are selected by the investigator to receive: Either Per the GORE Flow Reversal System IFU if the GORE Flow Reversal System is selected OR Per the GORE Embolic Filter IFU if the GORE Embolic Filter is selected

If the patient is contraindicated for both arms (devices) they may not be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1397 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - W.L. Gore and Associates, Inc, Flagstaff, Arizona
  - Hoag Memorial Hospital, Newport Beach, California
  - University of California San Francisco, San Francisco, California
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Kaiser FOundation Hospitals, Honolulu, Hawaii
  - Heart Care Research Foundation, Mokena, Illinois
  - Rockford Cardiovascular Associates, Rockford, Illinois
  - Indiana University, Indianapolis, Indiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Decaoness Medical Center, Boston, Massachusetts
  - Harper Hospital, Detroit, Michigan
  - St John's Medical Center, Detroit, Michigan
  - St Joseph Mercy Hospital, Pontiac, Michigan
  - Covenant Medical Center, Saginaw, Michigan
  - St Anthony's Medical Center, St Louis, Missouri
  - St Joesph's Medical Center, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Mercy Hospital, Buffalo, New York
  - Mt Sinai Hospital, New York, New York
  - St Francis Hospital, Roslyn, New York
  - Wake Heart Research, Raleigh, North Carolina
  - Forsyth Memorial Hospital, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - Heritage Valley Health Network, Beaver, Pennsylvania
  - Spirit Physician Services / Capital Cardiovascular Assoc, Camp Hill, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - N. Central Heart Hospital, Sioux Falls, South Dakota
  - St Luke's Episcopal, Houston, Texas
  - Appleton Medical Cetner, Appleton, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
  - St Lukes Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- GFRS EPD: Carotid artery stenting with Gore Flow Reversal System
  Gore Flow Reversal System: Embolic protection by the GORE Flow Reversal System during carotid artery angioplasty and stenting
- GEF EPD: Carotid artery stenting with Gore Embolic Filter
  Gore Embolic Filter: Embolic protection by the GORE Embolic Filter during carotid artery angioplasty and stenting
Period: Overall Study
Arm/Group | GFRS EPD | GEF EPD
Started | 425 | 972
Completed | 413 | 916
Not Completed | 12 | 56

BASELINE CHARACTERISTICS:
Population: All Enrolled Subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | GFRS EPD | GEF EPD | Total
Number analyzed (Participants) | 425 | 972 | 1397
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (8.7) | 73.0 (9.4) | 72.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 587 | 726
  Male | 286 | 385 | 671
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 16 | 27
  Not Hispanic or Latino | 414 | 955 | 1369
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants] — This measure is structured as a "check all that apply" field on the Case Report Form. Thus, the race categories are not mutually exclusive, except that "Not Reported" is mutually exclusive with the others. Because of this, the sum of the individual category counts is greater than the overall number of participants.
  participants
    American Indian or Alaska Native | 8 | 9 | 17
    Asian | 7 | 8 | 15
    Black or African American | 26 | 56 | 82
    Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
    White or Caucasian | 381 | 901 | 1282
    Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Events (MAE)
Description: Major Adverse Events include death, stroke and myocardial infarction
Time Frame: Onset from start of index procedure to 30-day follow-up assessment
Population: Enrolled subjects with successful procedure and sufficient follow-up
Measure: Number; unit: participants
Arm/Group | GFRS EPD | GEF EPD
Number analyzed (Participants) | 386 | 864
participants | 18 | 36

ADVERSE EVENTS:
Time Frame: 30-day visit window
Description: The Major Adverse Event components are reported as individual Serious Adverse Events. No other adverse events were collected in this study, so the number of subjects affected by Other (Not Including Serious) Adverse Events is zero (0).
Arm/Group | GFRS EPD | GEF EPD
Serious Adverse Events (participants affected / at risk) | 18/425 | 36/972
Other Adverse Events (participants affected / at risk) | 0/425 | 0/972
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFRS EPD (N=425) | GEF EPD (N=972)
All Cause Death (Cardiac disorders) | 2 (2) | 10 (10)
Myocardial Infarction (Cardiac disorders) | 6 (6) | 3 (3)
Stroke (Nervous system disorders) | 14 (14) | 31 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No